CLINICAL TRIAL: NCT03101878
Title: A Blinded, Placebo-Controlled, Dose-Escalation, Phase 1 Study to Assess the Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of Single and Multiple Doses of ISIS 757456 Administered Subcutaneously to Healthy Volunteers
Brief Title: Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of Ionis AGT-LRx in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Ionis Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ISIS 757456-CS1
Record Dates: First submitted 2017-03-06; First posted 2017-04-05 (Actual); Last update posted 2018-08-21 (Actual); Status verified 2018-08

CONDITIONS: Healthy Volunteers
Keywords: Healthy Volunteers, IONIS AGT-Lrx

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Ionis AGT-LRx (Experimental): Ascending single and multiple doses of Ionis AGT-LRx administered subcutaneously.
  Interventions: Drug: Ionis AGT-LRx
- Placebo (Placebo Comparator): Saline .9%
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Ionis AGT-LRx — Ascending single and multiple doses of Ionis AGT-LRx administered subcutaneously
  Arms: Ionis AGT-LRx
Drug: Placebo — Saline .9%
  Arms: Placebo

SUMMARY:
The purpose is to assess the Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of IONIS AGT-LRx in up to 82 Healthy Volunteers

ELIGIBILITY:
Inclusion Criteria:

* Must have given written informed consent and be able to comply with all study requirements
* Healthy males or females aged 18-60 inclusive and weighing ≥ 50 kg at the time of Informed Consent
* Females must be non-pregnant and non-lactating, and either surgically sterile or post- menopausal
* Males must be surgically sterile, abstinent or using an acceptable contraceptive method
* BMI ≤ 35 kg/m
* Agree to conduct at home blood pressure monitoring (in triplicate using study provided device) every morning and every evening throughout study participation for Single-Dose Cohort subjects and every morning for Multiple-Dose Cohort subjects

Exclusion Criteria:

* Treatment with another Study Drug, biological agent, or device within one-month of Screening
* Subject with borderline orthostatic hypotension defined as a fall in systolic blood pressure of ≥ 17 mmHg or diastolic blood pressure of ≥ 7 mmHg when they assume a standing position (within 3 minutes of standing up)
* Use of nicotine-containing products or illicit drugs
* Considered unsuitable for inclusion by the Principal Investigator

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 62 (Actual)
Dates: Start 2017-04-05 (Actual); Primary Completion 2018-03-29 (Actual); Study Completion 2018-08-01 (Actual)

PRIMARY OUTCOMES:
Incidence and severity of adverse events that are related to treatment with IONIS AGT-LRx | Up to 127 days
  The safety and tolerability of single and multiple doses of IONIS AGT-LRx will be assessed by determining the incidence, severity, and dose relationship of adverse events that are related to treatment with IONIS AGT-LRx
Any observed changes in Blood Pressure measurements, ECGs, or laboratory tests from baseline | Up to 127 days
  The safety and tolerability of single and multiple doses of IONIS AGT-LRx will be assessed by reviewing any observed changes in Blood Pressure measurements, physical exam, and laboratory tests from baseline by dose. Results in subjects dosed with IONIS AGT-LRx will be compared with those from subjects dosed with placebo.

SECONDARY OUTCOMES:
Pharmacokinetics after single and multiple doses of IONIS AGT-LRx | Up to 127 days
  The plasma pharmacokinetics (concentration-time results) of IONIS AGT-LRx will be assessed following single and multiple dose SC administration
Pharmacodynamics of IONIS AGT-LRx (Changes in plasma AGT Levels) | Up to 127 days
  Effects of IONIS AGT-LRx on changes in AGT plasma protein compared to baseline.

CONTACTS AND LOCATIONS:
Locations (1):
- Syneos Health, Toronto, Ontario, Canada

REFERENCES:
- [Derived] Morgan ES, Tami Y, Hu K, Brambatti M, Mullick AE, Geary RS, Bakris GL, Tsimikas S. Antisense Inhibition of Angiotensinogen With IONIS-AGT-LRx: Results of Phase 1 and Phase 2 Studies. JACC Basic Transl Sci. 2021 May 3;6(6):485-496. doi: 10.1016/j.jacbts.2021.04.004. eCollection 2021 Jun. PMID 34222719